CLINICAL TRIAL: NCT04837014
Title: Eliminating Narcotic Prescriptions from Outpatient Minimally Invasive Gynecologic Surgery: a Randomized Controlled Trial
Brief Title: Eliminating Narcotic Prescriptions from Outpatient Minimally Invasive Gynecologic Surgery
Acronym: eNARCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Andrew Zakhari, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F11-70846
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative; Opioid Use
Keywords: Gynecology; Minimally invasive surgery; Laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Prescriptions; Naproxen; Hydromorphone

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, consented patient will be randomly allocated to either intervention or control groups in a 1:1 fashion. Allocation will be determined by a computerized randomization generator with block randomization in groups of four. Allocations will be placed in sequentially numbered, sealed, opaque envelopes to be opened only upon completion of surgery of consenting patients.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Although the patient and operative team will not be blinded to the allocation, the research team member completing the post-operative questionnaires as well as the statistician responsible for data analysis will remain blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen and naproxen only arm (Experimental): Patient allocated to the intervention arm will be discharged home with a prescription for regular acetaminophen and naproxen for 48 hours, and then as needed for one week's duration.
  Interventions: Other: prescription for regular acetaminophen and naproxen
- Acetaminophen, naproxen and dilaudid arm (Active Comparator): Patient allocated to the control group will be discharged home with a prescription for regular acetaminophen, naproxen, and 5 tabs of hydromorphone 1 mg, with instruction to prioritize non opioid analgesic as first line.
  Interventions: Other: prescription for regular acetaminophen , naproxen and dilaudid

INTERVENTIONS:
Other: prescription for regular acetaminophen and naproxen — Patient allocated to the intervention arm will be discharged home with a prescription for regular acetaminophen and naproxen for 48 hours, and then prn for one week's duration. No narcotic will be prescribed at discharge post-operatively.
  Arms: Acetaminophen and naproxen only arm
Other: prescription for regular acetaminophen , naproxen and dilaudid — prescription for regular acetaminophen , naproxen and dilaudid
  Arms: Acetaminophen, naproxen and dilaudid arm

SUMMARY:
Laparoscopic gynecologic surgeries are generally very well tolerated procedures, and patients are able to go home on the same day, with a prescription for pain control. There is currently a very wide range of prescription practice within the gynecology community in regards to opioids following surgery, and patients are going home with anything from zero to 5 or even 20 tabs of narcotics.

Aside from negative side effect of opioids (like nausea/vomiting, dizziness, constipation, and possibly addiction), unnecessary opioid prescriptions and excess unused narcotics is one of the major contributors to narcotic abuse in the community, worsening an ongoing nationwide opioid crisis. Although most patients report low pain level following these kinds of procedure, there are no current standard prescriptions after gynecologic laparoscopy.

In an effort to standardize discharge prescriptions following gynecologic laparoscopy, this study aims to find an optimal regimen for pain control in the post-operative period following laparoscopic gynecologic surgery. There will be 2 standardized set of discharge prescriptions to which patient will be randomized; both containing multimodal medications for pain control. Pain control, and patients satisfaction will be measured in the first post-operative week.

DETAILED DESCRIPTION:
Narcotic prescribing patterns vary greatly among gynecologists performing minimally invasive gynecologic surgery (MIGS). There is no clear consensus or established guideline regarding the choice of narcotic or total amount to be prescribed, if any, for MIGS. These represent a generally well-tolerated group of procedures that are less painful than conventional open surgery. Unnecessary opioid prescriptions and excess unused narcotics have been identified as major contributors to narcotic abuse in the community, and efforts geared towards minimizing unnecessary narcotic prescriptions may help curb the growing opioid crisis.

This study suggests eliminating opioids from discharge prescriptions following outpatient MIGS in select patients. Given the general tolerability and low pain associated with MIGS, the investigators hypothesize that elimination of narcotics from post-operative pain control, in conjunction with regular use of non-narcotic analgesics, will result in analgesia and early recovery that is no worse than a standard narcotic-containing discharge prescription.

Women undergoing elective outpatient laparoscopic gynecologic surgery at two medical center associated with the McGill University Health Centre will be recruited and screened for exclusion criteria. Patients will be randomly allocated to either intervention or control groups in a one to one fashion. Patients in both intervention and control group will undergo surgery under a standardized anesthesia protocol. Important surgical steps that can affect post-operative pain will be standardised and recorded with a surgical checklist to reduce inter-surgeon variability. Patient allocated to the intervention arm will then be discharged home with a prescription for regular acetaminophen and naproxen for 48 hours, and then as needed for one week's duration. Patient in control group will be discharge with a standard prescription of five tabs of 1 mg hydromorphone, with regular non-opioid analgesic use.

All patient will be contacted on day one and seven after surgery to evaluate pain scores, mobility, adequacy of analgesia, adherence to treatment, side-effects, and total opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective outpatient gynecologic laparoscopy
* Able to provide informed consent
* Planned for same day discharge

Exclusion Criteria:

* Chronic pain conditions including, but not limited to: chronic pelvic pain, fibromyalgia, connective tissue disorders, migraines on medication, severe osteoarthritis, sciatica, degenerative disk disease
* Regular use of analgesia or narcotics. Defined as use of pain medication on most days of the week, most weeks of the month
* History of substance abuse (opioid addiction, IV drug use, etc.)
* Known depression or anxiety conditions with or without medication
* Eastern Cooperative Oncology Group (ECOG) performance status 3 or greater
* Current or recent use of pain modulators such as pregabalin or gabapentin (one month pre-operatively).
* Allergy or contraindication to acetaminophen or NSAIDs or hydromorphone/narcotics
* Intraoperative complications :
* Conversion to laparotomy or mini-laparotomy > 4 cm
* Intra-operative gastrointestinal or urologic injury
* Intra-operative hemorrhage or need for blood transfusion
* Need for admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Pain score on post-operative day one | Post-operative day one
  The primary outcome of this study is patient reported pain using an 11-point Numerical Rating Scale (NRS) on post-operative day two, on a scale from 0 to 10 in which higher scores indicate higher pain (worse pain control).

SECONDARY OUTCOMES:
Patient mobility and satisfaction of analgesia | Post-operative day one and seven
  Patients will receive a phone call on post-operative day one and seven and will be asked a standardised set of questions binary question (Yes / No) to evaluate patient mobility and satisfaction of analgesia.
Total narcotic consumption in the first post-operative week | Post-operative day seven
  Patients will receive a phone call on post-operative day one and seven and will be asked total amount of narcotic consumed since discharge from the hospital, including need for rescue prescription
Opioid related side effect | First post-operative week (Day 7)
  Patients will receive a phone call on post-operative day one and seven and will be inquired about specific opioid side effect.
Unplanned return to emergency room / clinic | First post-operative week (Day 7)
  Patients will receive a phone call on post-operative day one and seven and will be inquired about any unplanned visit to emergency room / clinic since discharged from the hospital.
Overall satisfaction with pain control | First post-operative week (Day 7)
  Patients will receive a phone call on post-operative day one and seven and will be asked about overall satisfaction with pain control via standardised questionnaire.
Pain score on post-operative day one | Post-operative day 7
  Patient reported pain using an 11-point Numerical Rating Scale (NRS) on post-operative day one, on a scale from 0 to 10 in which higher scores indicate higher pain (worse pain control).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zakhari, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zakhari A, Desilets J, Della Rocca C, Shan WLP, Nguyen DB, Gilbert L, Smith JP, Krishnamurthy S, Mansour FW. Eliminating opioid prescriptions from outpatient minimally invasive gynecologic surgery: a randomized trial. Nat Med. 2026 Jan 5. doi: 10.1038/s41591-025-04096-6. Online ahead of print. PMID 41491106